CLINICAL TRIAL: NCT00445094
Title: A De-Escalating Strategy for Antibiotic Treatment of Pneumonia in The Medical Intensive Care Unit
Brief Title: A De-Escalating Strategy for Antibiotic Treatment of Pneumonia in The Medical Intensive Care Unit (0787B-092)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0787B-092; 2007_004
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Infection; Pneumonia
MeSH Terms: conditions — Infections; Pneumonia | interventions — Imipenem; Cilastatin; Duration of Therapy

INTERVENTIONS:
Drug: MK0787B, imipenem/cilastatin sodium / Duration of Treatment: 7 Days
Drug: Comparator: amikacin / Duration of Treatment: 3 Days
Drug: Comparator: tazocin / Duration of Treatment: 3 Days
Drug: Comparator: vancomycin / Duration of Treatment: 3 Days

SUMMARY:
The primary objective of this study is a comparison between MK0787B and standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Patient is diagnosed with nosocomial pneumonia

Exclusion Criteria:

* Immunological deficient patients
* Pregnant women and nursing mothers
* A fungus is identified before the study enrollment
* Received vancomycin or imipenem for more than 5 days before icu admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
A 30-day-survival rate in the intensive care unit evaluated by Acute Physiology and Chronic Health (APACH II) Disease Classification System II score

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html